CLINICAL TRIAL: NCT01755312
Title: The Effect of Medication Reminder Technology on Medication Adherence and Hypertension
Brief Title: The Effect of Medication Reminder Technology on Medication Adherence and Hypertension Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research site no longer available
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Alan Zillich Lab, Associate Professor Pharmacy Practice, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2r44ago39178-02 (1208012596)
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Medication Adherence; Blood Pressure
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- medication reminder (Experimental): medication reminder
  Interventions: Device: Medication reminder
- Placebo (Placebo Comparator): Placebo

INTERVENTIONS:
Device: Medication reminder — Medication reminder
  Arms: medication reminder

SUMMARY:
This study to evaluates how a med reminder affects the patient's ability to take medications as prescribed

ELIGIBILITY:
Inclusion Criteria:

* poor medication adherence
* high blood pressure

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
self-reported medication adherence using the Morisky 8-Item Medication Adherence Scale(MMAS-8) tool | 6 months

SECONDARY OUTCOMES:
systolic blood pressure in mmHg using a valid automated device | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States